CLINICAL TRIAL: NCT05985629
Title: The Effect of IPACK Nerve Blocks on Early ACL Pain Scores
Brief Title: IPACK on Early Pain Scores After ACL Reconstruction
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LU 216180
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Pain, Postoperative; Anterior Cruciate Ligament Injuries; Analgesics, Opioid
MeSH Terms: conditions — Pain, Postoperative; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: An unblinded pharmacist will prepare the study drugs consisting of IPACK block, or the sham block consisting of saline (control group). All patients will be premedicated with midazolam, which is standard of care prior to general anesthesia. The use of a sham block, administered by the anesthesia team, is to ensure that the Investigator is blinded to patient's treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IPACK (Experimental): After the adductor canal block, the anesthesiologist will reposition, visualize the anatomy of the IPACK block with ultrasound, and place 1% lidocaine for skin infiltration. Once adequate needle visualization is achieved within the correct anatomic position and plane, 20mL of 0.5% bupivacaine will be injected.
  Interventions: Drug: IPACK
- Placebo (Placebo Comparator): After the adductor canal block, the anesthesiologist will reposition, visualize the anatomy of the IPACK block with ultrasound, and place 1% lidocaine for skin infiltration. Once adequate needle visualization is achieved within the correct anatomic position and plane, 20mL of normal saline will be injected.
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: IPACK — Infiltration between the popliteal artery and capsules of the knee (IPACK) is a novel ultrasound-guided technique that provides additional regional analgesic relief to the posterior aspect of the knee without complications seen in a sciatic nerve block. The intention of the IPACK block is to anesthetize the terminal sensory nerves while sparing the main trucks of the common peroneal and tibial nerves.
  Arms: IPACK
Drug: PLACEBO — The control group will receive the normal pre-procedure care including a pre-operative visit, surgery, and post-operative care. The control group will receive a sham block consisting of saline in the same anatomical location and manner that the intervention IPACK block is administered.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn whether using an anesthetic technique called IPACK block will control pain after ACL reconstruction surgery. The main questions it aims to answer are:

* if participants who receive the IPACK block prior to ACL reconstruction experience less pain after surgery and at 1 day after surgery
* if participants who receive the IPACK block prior to ACL reconstruction require less short-term opioid use immediately after surgery and up to one week after surgery.

Participants will be randomized 1:1 to 1 of 2 groups: Use of IPACK block during ACL reconstruction vs. placebo (a placebo is a look-alike substance that contains no active drug). Neither the participant nor the investigator will know which group the participants has been assigned to.

Researchers will compare self-reported pain scores and short-term opioid use of all study participants.

DETAILED DESCRIPTION:
Eligible patients will be approached for voluntary study participation after they have made the decision to pursue an elective ACL reconstruction surgery with Dr. John Miller of Loyola University Department of Orthopedic Surgery for management of their ACL tear.

The study design is a double-blind, randomized trial. Patients will be randomly selected to the control group or the treatment group. The groups will be randomized 1:1 using a block method to be implemented. The control group will receive a sham block, while the treatment group will receive the IPACK block. The use of a sham block, administered by the anesthesia team, is to ensure that Dr. Miller is blinded to patient's treatment group. After administration of the block and a completed ACL reconstruction surgery, pain scores will be collected from the patient at two time points. First, pain scores will be collected in the post-anesthesia care (PACU) unit using the visual analogue scale (VAS) immediately upon waking up, one hour after waking up and upon discharge. Second, pain scores will be collected during the standard post-operative follow-up phone call that Dr. Miller makes with all his patients one day after surgery using the VAS pain scale. Short-term postoperative opioid consumption will be measured in the PACU by calculating the milligram-equivalents of morphine used by patients' starting at their arrival until their discharge. This data will be extracted from the patient's chart on EPIC. Information about the patient's opioid use from discharge until 1-week post-operatively will be collected either in person at the patient's first outpatient post-operative follow up or via patient phone call one week after surgery using a simple questionnaire

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to Dr. John Miller with the Department of Orthopedic Surgery, Sports Medicine Division, at Loyola University Medical Center electing to undergo ACL reconstruction surgery.
* Patients 16 and over
* English speaking patients
* Patients who have the capacity to make their own medical decisions and consent to the study

Exclusion Criteria:

* Previous surgery on the operative knee
* Previous knee infection
* Chronic opioid use
* Have a known allergy to local anesthetics
* Patient using autograft (cadaver) for ACL reconstruction.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-08-03 (Estimated); Study Completion 2026-08-03 (Estimated)

PRIMARY OUTCOMES:
Pain Scores | Immediately after surgery; 1 hour, 2-3 hours, and 24 hours after surgery
  Visual Analogue Scale (VAS). Participants self-report their post surgical pain from a scale of 0 to 10.
Opioid Consumption | 2-3 hours after surgery; 1 week after surgery
  Short-term postoperative opioid consumption will be measured in the PACU by calculating the milligram-equivalents of morphine used by patients' starting at their arrival until their discharge. This data will be extracted from the patient's chart on EPIC. Information about the patient's opioid use from discharge until 1-week post-operatively will be collected either in person at the patient's first outpatient post-operative follow up or via patient phone call one week after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do not have intentions on sharing IPD with other researchers at this time. If we decide to collaborate in the future, IPD will be de-identified prior to sharing.

REFERENCES:
- Available data/document: Study Protocol — https://hsd.luc.edu/cro/ — Information about this study can be requested from the Clinical Research Office at Loyola University Chicago by calling 708-216-1153 or by mail at: Loyola University Chicago Center for Translational Research and Education (CTRE) Bldg. 115, Suite 253, Rm 255 Maywood, IL 60153